CLINICAL TRIAL: NCT00025649
Title: European Infant Neuroblastoma Study - Stage 2, 3, 4, and 4S; MYCN Amplified Tumors
Brief Title: Combination Chemotherapy Followed by Surgery and Peripheral Stem Cell or Bone Marrow Transplantation in Treating Infants With Newly Diagnosed Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Infant Neuroblastoma Study Group - 1999 (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068982; EURO-INF-NB-STUDY-1999-99.4; EU-20125D
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2001-12

CONDITIONS: Neuroblastoma
Keywords: localized resectable neuroblastoma; regional neuroblastoma; disseminated neuroblastoma; stage 4S neuroblastoma; localized unresectable neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; Busulfan; Carboplatin; Cyclophosphamide; Doxorubicin; Etoposide; Melphalan; Vincristine; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: busulfan
Drug: carboplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: melphalan
Drug: vincristine sulfate
Procedure: autologous bone marrow transplantation
Procedure: conventional surgery
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell or bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy given before surgery followed by peripheral stem cell or bone marrow transplantation in treating infants who have newly diagnosed neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the survival of infants with newly diagnosed stage II, III, IV, or IVS neuroblastoma with MYCN amplification treated with etoposide, carboplatin, cyclophosphamide, doxorubicin, and vincristine followed by surgery and busulfan and melphalan with autologous peripheral blood stem cell or bone marrow transplantation.
* Determine whether there are prognostic criteria that could be used in future therapeutic stratification of these patients.

OUTLINE: This is a multicenter study.

Patients receive VP-CARBO chemotherapy comprising etoposide IV over 2 hours and carboplatin IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 courses. Patients then receive CADO chemotherapy comprising cyclophosphamide IV over 1 hour on days 1-5, doxorubicin IV over 6 hours on days 4 and 5, and vincristine IV on days 1 and 5. Treatment repeats every 21 days for 2 courses.

Patients receive filgrastim (G-CSF) subcutaneously daily for 5 days. Patients undergo leukapheresis to collect peripheral blood stem cells (PBSC). Patients who do not mobilize sufficient cells undergo bone marrow harvest.

Patients eligible for surgery undergo surgical resection. Patients with stage IV disease with less than complete response of metastatic disease after initial chemotherapy are removed from the study.

Beginning within 2 weeks after surgery, patients receive 1 additional course of VP-CARBO chemotherapy followed by 1 additional course of CADO chemotherapy.

After at least 3 weeks, patients receive high-dose chemotherapy comprising busulfan IV over 24 hours on days -7 to -3 and melphalan IV on day -2. PBSC or bone marrow are reinfused on day 0.

At least 2 months after the completion of high-dose chemotherapy and bone marrow or PBSC transplantation, patients undergo radiotherapy to the primary site, according to preoperative imaging studies. Patients are treated with oral tretinoin after megatherapy.

Patients are followed within 6 months and then annually for 5 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed stage II, III, IV, or IVS neuroblastoma or ganglioneuroblastoma
* MYCN amplification (i.e., at least 10 copies)

PATIENT CHARACTERISTICS:

Age:

* Under 12 months at diagnosis

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1999-07; Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adela Canete, MD, PhD, Study Chair — Hospital Universitario La Fe
Locations (11):
- St. Anna Children's Hospital, Vienna, Austria
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Rigshospitalet, Copenhagen, Denmark
- Centre Hospitalier Regional de Purpan, Toulouse, France
- Istituto Giannina Gaslini, Genoa, Italy
- Rikshospitalet University Hospital, Oslo, Norway
- Instituto Portugues de Oncologia de Francisco Gentil - Centro Regional de Oncologia de Lisboa, S.A., Lisbon, Portugal
- Hospital Universitario LA FE, Valencia, Spain
- Ostra Sjukhuset, Gothenburg, Sweden
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- Bristol Royal Hospital for Children, Bristol, England, United Kingdom

REFERENCES:
- [Result] Canete A, Gerrard M, Rubie H, Castel V, Di Cataldo A, Munzer C, Ladenstein R, Brichard B, Bermudez JD, Couturier J, de Bernardi B, Pearson AJ, Michon J. Poor survival for infants with MYCN-amplified metastatic neuroblastoma despite intensified treatment: the International Society of Paediatric Oncology European Neuroblastoma Experience. J Clin Oncol. 2009 Mar 1;27(7):1014-9. doi: 10.1200/JCO.2007.14.5839. Epub 2009 Jan 26. PMID 19171715